CLINICAL TRIAL: NCT06035250
Title: Deep Learning-Based Prediction of Gastric Cancer Response to Neoadjuvant Chemotherapy
Brief Title: AI Prediction of Gastric Cancer Response to Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Yunnan Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Zhenjiang First People's Hospital (Other); First Hospital of China Medical University (Other); Cancer Hospital of Guangxi Medical University (Other); Peking University People's Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Nanfang Hospital, Southern Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Ruijin Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking Union Medical College Hospital (Other); Xiangya Hospital of Central South University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); The First Affiliated Hospital of Soochow University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Fujian Medical University Union Hospital (Other); Fujian Cancer Hospital (Other Government); San Raffaele University Hospital, Italy (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Institute of Automation, Chinese Academy of Sciences
Other Study IDs: CASMI004
Record Dates: First submitted 2023-08-13; First posted 2023-09-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; Image; Pathology
Keywords: Gastric Cancer; Neoadjuvant Chemotherapy; Radiomics; Treatment Outcome Prediction; Pathomics; Radiopathomics
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biospecimens consist of gastric tumor biopsy samples, collected from each patient prior to the initiation of neoadjuvant chemotherapy. These specimens undergo HE (Hematoxylin and Eosin) staining for pathology imaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric Cancer Patients Undergoing Neoadjuvant Chemotherapy: This group comprises participants diagnosed with advanced gastric cancer. The participants will be treated with standard neoadjuvant chemotherapy regimens recommended by clinical guidelines. Treatment details, including the generic name of the drugs, dosage form, dosage, frequency, and duration, will be recorded according to the specific regimen.
  Interventions: Drug: Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — Participants in this group are diagnosed with gastric cancer and are scheduled to undergo neoadjuvant chemotherapy as a part of their treatment regimen. The specific chemotherapy drugs, dosages, and schedules will be determined according to established clinical guidelines and the participant's specific condition.

SUMMARY:
This study seeks to develop a deep-learning-based intelligent predictive model for the efficacy of neoadjuvant chemotherapy in gastric cancer patients. By utilizing the patients' CT imaging data, biopsy pathology images, and clinical information, the intelligent model will predict the post-neoadjuvant chemotherapy efficacy and prognosis, offering assistance in personalized treatment decisions for gastric cancer patients.

DETAILED DESCRIPTION:
This study seeks to develop a deep learning model to predict the outcomes of neoadjuvant chemotherapy in patients with gastric cancer. Leveraging participants' CT scans, biopsy pathology images, and clinical profiles, this model aims to forecast the effectiveness of post-neoadjuvant chemotherapy and the subsequent prognosis, thereby aiding in individualized treatment choices for these participants.

Data Collection: The investigators will gather data from 1,800 retrospective cases and 200 prospective cases from multiple hospitals. The retrospective data will be divided into training and testing sets to train and validate the model, respectively. The model's performance will subsequently be evaluated using the prospective dataset.

Clinical Information: This encompasses the participant's gender, age, tumor markers, staging, type, specific treatment plans, pre and post-treatment lab results, etc.

Imaging Data: CT imaging data taken within one month prior to the neoadjuvant chemotherapy, with at least the venous phase CT imaging included.

Pathology Data: Pathology images from a gastric tumor biopsy stained with Hematoxylin and Eosin (HE) taken within one month prior to treatment.

TRG Grading: Based on the pathology report of the surgical samples using the Ryan TRG grading system.

Prognostic Endpoints: The recorded endpoints are a 3-year progression-free survival (PFS) and a 5-year overall survival (OS). All deaths due to non-disease factors are excluded from the prognosis analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Pathologically diagnosed with advanced gastric cancer in accordance with the American AJCC's TNM staging standards;
* Have not undergone any systematic anti-cancer treatments before neoadjuvant chemotherapy and have not had surgery for local progression or distant metastasis;
* Received standard neoadjuvant chemotherapy as recommended by the clinical guidelines, and have documented treatment details;
* CT imaging and biopsy pathology images strictly taken within one month prior to starting neoadjuvant treatment;
* Patients possess comprehensive preoperative clinical information and post-operative TRG grading.

Exclusion Criteria:

* Patients whose CT or pathology images are unclear, making lesion assessment infeasible;
* Patients diagnosed with other concurrent tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises gastric cancer patients from various hospitals. Participants are individuals diagnosed with advanced gastric cancer and are currently undergoing neoadjuvant chemotherapy treatments. Selection is based on criteria such as age, specific diagnosis, past treatment history, and the clarity of their medical images and pathology images.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC) for TRG prediction by the AI model | two months
  The AUC will be used to evaluate the performance of the AI model in predicting TRG grading of gastric cancer patients after neoadjuvant chemotherapy. An AUC of 1 indicates perfect prediction, while an AUC of 0.5 indicates prediction no better than chance.
Accuracy of TRG prediction by the AI model | two months
  Accuracy measures the proportion of true positive and true negative predictions made by the AI model among all predictions. It indicates the capability of the model to correctly classify patients into their respective TRG gradings.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) at 3 years | Three years
  The duration from the date of patient confirmation to the date of tumor progression or death of the patient, whichever occurs first.
Overall Survival (OS) at 5 years | Five years
  The duration from the date of patient confirmation to the date of death of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yali Zang, Ph.D., Study Director — Institute of Automation, Chinese Academy of Sciences
Locations (22):
- China (21):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Cancer Hospital & Institute, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Yunnan Cancer Hospital, Kunming
  - Cancer Hospital of Guangxi Medical University, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Ruijin Hospital, Shanghai
  - First Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhenjiang First People's Hospital, Zhenjiang
- San Raffaele University Hospital, Italy, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) may be made available to other researchers upon request. Interested researchers should present a reasonable research proposal and a data usage application. All participating units of this study will review and assess the proposal and application to determine whether to share the data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available 1 year after study completion and will remain available for a period of 5 years.
Access Criteria: Interested researchers should submit a detailed research proposal and a data usage application for review. All participating units of this study will assess the application to determine eligibility for data access.
URL: http://www.radiomics.net.cn/